CLINICAL TRIAL: NCT05570253
Title: "A Phase 2, Double Blinded, Randomized Controlled Trial of Evexomostat (SDX-7320) or Placebo in Combination With Eribulin for Patients With Metastatic Triple-Negative Breast Cancer and Metabolic Dysfunction: The ARETHA Study
Brief Title: A Study of SDX-7320 in Combination With Eribulin for People With Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: SynDevRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-074
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; Metastatic Triple-Negative Breast Cancer
Keywords: Evexomostat (SDX-7320); Eribulin; 22-074
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Intervention Model Description: This is a multi-center, placebo-controlled phase 2 randomized control trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SDX-7320 plus Eribulin (safety run-in period) (Experimental): During the safety run-in period, the first 15 patients enrolled will be assigned to received study drug SDX-7320 plus Eribulin. Not randomized.
  Interventions: Drug: Eribulin; Drug: SDX-7320
- SDX-7320 plus Eribulin (Experimental): Patients randomized to SDX-7320 plus Eribulin.
  Interventions: Drug: Eribulin; Drug: SDX-7320
- Eribulin Plus Placebo (Placebo Comparator): Patients randomized to the control arm will receive placebo plus Eribulin.
  Interventions: Drug: Eribulin; Other: Placebo

INTERVENTIONS:
Drug: Eribulin — Eribulin 1.4 mg/m2 IV on days 1 and 8 of an every 21 day cycle.
Drug: SDX-7320 — SDX-7320 at the dose of 49 mg/m2 SC on a Q14D basis
  Arms: SDX-7320 plus Eribulin; SDX-7320 plus Eribulin (safety run-in period)
Other: Placebo — Placebo
  Arms: Eribulin Plus Placebo

SUMMARY:
The researchers are doing this study to find out whether the study drug, SDX-7320, when combined with the standard chemotherapy eribulin, is an effective treatment for people with TNBC and metabolic dysfunction. The researchers will also look at whether the study treatment (SDX-7320 combined with eribulin) is safe and causes few or mild side effects in participants. The researchers will compare this treatment approach to eribulin alone.

DETAILED DESCRIPTION:
The study includes a safety run-in period in which the first 15 patients enrolled will be assigned to receive the study drug SDX-7320 in combination with eribulin. Upon safety confirmation, randomization will commence for the subsequent 40 patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with histologically and/or cytologically confirmed diagnosis of triple-negative metastatic breast cancer defined as estrogen and progesterone receptor staining ≤10%; and HER2-negative defined as IHC 0 to 1+ at enrolling institution (note: if IHC is equivocal, non-amplified status by FISH is acceptable)
* Advanced (local regionally recurrent, not amenable to curative therapy or surgery) or metastatic stage with up to 2 prior lines of therapy in the advanced or metastatic setting
* Received prior anthracycline and taxane chemotherapy in the neoadjuvant, adjuvant, or metastatic settings and considered appropriate for treatment with single agent eribulin OR was otherwise ineligible to receive anthracycline and/or taxane per treating physician OR patients with de novo metastatic disease.
* Evidence of metabolic dysfunction defined as HbA1c > 5.5 and/or BMI ≥ 30 kg/m^2
* Measurable disease per the Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1), OR at least one evaluable, predominantly lytic bone lesion
* Eastern Cooperative Oncology Group Performance Status (ECOG-PS) ≤1.
* Adult ≥18 at the time of informed consent and has provided written informed consent before the performance of any study-related activities and according to local guidelines.
* Adequate bone marrow and organ function as defined by the following laboratory values (as assessed by local laboratory for eligibility):

  * Absolute neutrophil count (ANC) ≥ 1,000 µL
  * Platelet count ≥ 140,000 µL
  * Hemoglobin ≥9.0 g/dL:
  * Calcium (corrected for serum albumin) and magnesium ≤ Grade 1 according to National Cancer Institute (NCI) Common Terminology
  * Calculate Corrected Calcium if the albumin and/or serum calcium are not within normal limits: Corrected Calcium= Serum Calcium + 0.8 x [(Normal Albumin) - Patient Albumin] Normal Albumin value = 4.4g/dL Criteria for Adverse Events (CTCAE), version 5.0, and not considered by the Investigator to be clinically significant
  * Potassium within normal limits, with or without correction with supplements.
  * In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×the upper limit of normal (ULN). If the patient has liver metastases, ALT and AST ≤5×ULN.
  * Total bilirubin ≤1.5×ULN except for patient with Gilbert's syndrome who may only be included if the total bilirubin is ≤3.0×ULN or direct bilirubin ≤1.5×ULN
  * Creatinine ≤1.5 mg/dL.
* Patient is, in the treating Investigator's opinion, willing and able to comply with the study requirements, including the ability to fast prior to treatment days.
* If sexually active female of childbearing potential, willing to use a contraception method listed below:

  * Oral, intravaginal, or transdermal combined (estrogen and progesterone containing) hormonal contraception
  * Oral, injectable, or implantable progesterone-only hormonal contraception
  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomized partner with documentation of successful vasectomy.
  * Complete abstinence from heterosexual intercourse
* If a sexually active male, willing to use barrier contraception (condoms)

Exclusion Criteria:

* Three or greater prior lines of therapy for metastatic TNBC
* Known primary brain malignancy, brain metastases or active CNS pathology, any of which as determined by the treating Investigator
* Currently participating in a study of an investigational agent
* Body mass index < 18.5 kg/m2
* Known hypersensitivity to SDX-7320 or eribulin
* Established diagnosis of diabetes mellitus type I or uncontrolled or insulin-dependent type II. Uncontrolled is defined as fasting blood glucose >140 mg/dL and/or HbA1c ≥8%
* Use of combination antihyperglycemic therapy (single agent metformin on stable dose for at least 3 months prior to enrollment is allowable)
* Concurrent malignancy or malignancy within 3 years of randomization, with the exception of adequately treated, basal or squamous cell carcinoma, nonmelanomatous skin cancer or curatively resected cervical cancer.
* Uncontrolled human immunodeficiency virus (HIV) infection. (Testing is not mandatory.)
* Evidence of uncontrolled active Hepatitis B or C infection
* History of Stevens-Johnson Syndrome (SJS), erythema multiforme (EM), toxic epidermal necrolysis (TEN), or other severe medication-related cutaneous reactions.
* Any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment, contraindicate patient participation in the clinical study (e.g., chronic active hepatitis, severe hepatic impairment).
* Clinically significant, uncontrolled heart disease and/or recent cardiac events including any of the following:

  * History of angina pectoris, coronary artery bypass graft (CABG) symptomatic pericarditis, or myocardial infarction within 6 months prior to study entry.
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV).
  * Documented cardiomyopathy.
  * Left ventricular ejection fraction (LVEF) <45%, as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO).
  * History of any cardiac arrhythmias, (e.g., ventricular tachycardia), complete left bundle block, high grade atrioventricular (AV) block (e.g., bifascicular block, Mobitz type II and third-degree AV block) supraventricular, nodal arrhythmias, or conduction abnormality in the previous 12 months.
  * Uncontrolled hypertension, defined by a systolic blood pressure (SBP) ≥160 mmHg and/or diastolic blood pressure (DBP) ≥100 mmHg, with or without antihypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening
  * Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome or any of the following: risk factors for torsades de pointe including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure or history of clinically significant/symptomatic bradycardia; concomitant medications with a known risk to prolong the QT interval and known to cause torsades de pointe that cannot be discontinued or replaced by safe alternative medications.
  * Bradycardia (heart rate less than 50 at rest), by electrocardiogram (ECG) or pulse.
  * Inability to determine the QT interval on the ECG (i.e., unreadable or not interpretable) or corrected QT (QTcF) >450 msec for males and >470 msec for females (using Fridericia's correction) during Screening, based on the mean of triplicate ECGs
* Currently receiving any of the following medications and cannot be discontinued 7 days prior to the start of the treatment: Medications with a known risk to prolong the QT interval or induce Torsade de Pointes (TdP). CredibleMeds list of drugs known to cause TdP may be used as a reference for this study to determine which drugs are prohibited using the following link: https://crediblemeds.org/new-drug-list or a crediblemeds mobile application.

  °Herbal preparations/medications, with the exception of cannabinoids, CBD compounds, etc.
* Participation in a prior investigational study within 14 days prior to the start of the study treatment or within 5 half-lives of study drug, whichever is longer.
* History of acute pancreatitis within 1 year of Screening or past medical history of chronic pancreatitis
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
change in insulin resistance scores (HOMA-IR) | 1 year
  The Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) is a validated tool for the assessment of insulin resistance.87 HOMA-IR is calculated as follows: fasting serum insulin (μU/mL) × fasting plasma glucose (mmol L
  -1 )/22.5).

SECONDARY OUTCOMES:
Type, frequency and severity of treatment-emergent adverse events | 2 years
  (TEAEs) and laboratory toxicities per the NCI CTCAE version 5.0.
Overall response rate | 1 year
  Response rate will be assessed by RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Shen, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - BAPTIST ALLIANCE - MCI (Data Collection Only), Miami, Florida
  - Emory University (Data Collection Only), Atlanta, Georgia
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm